CLINICAL TRIAL: NCT06248450
Title: Medical Yoga During Cancer Treatment in a Digital or Physical Setting - a Preference-based Study
Brief Title: Medical YOga dUring CANcer Treatment in a Digital or Physical Setting - a PREFERensbased Study
Acronym: YouCanPrefer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: University Hospital, Linkoeping (Other); Ryhov County Hospital (Other)
Responsible Party: Principal Investigator, Anna Stroemberg, professor, Linkoeping University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-04481-01
Record Dates: First submitted 2024-01-07; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Cancer
Keywords: oncological treatment; yoga; e-health; rehabilitation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Preference-based allociation to group yoga in a physical or in a digital setting
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical setting (Other): Medical yoga at a yoga local led by a yoga-instructor for 75 minutes once a week and individual yoga for a minimum of 10 minutes daily using a yoga-application for 12 weeks.
  Interventions: Other: Medical yoga
- Digital setting (Other): Medical yoga online using videoconference system led by a yoga-instructor for 75 minutes once a week and individual yoga for a minimum of 10 minutes daily using a yoga-application for 12 weeks.
  Interventions: Other: Medical yoga

INTERVENTIONS:
Other: Medical yoga — Medical yoga is a therapeutic form of Kundalini yoga led by a certified yoga instructor that uses different standardized yoga programs with a combination of physical postures, breathingexercises, and relaxation/meditation.

SUMMARY:
To enhance the implementation of yoga in cancer care, studies that explore patients with cancer preferences for the execution of yoga, effects, and the experience of participating in group yoga sessions online compared to in-person sessions is required. The aim of the YouCanPrefer-study is to explore preferences, expectations, implementation, experiences, and effects of participating in in-person group yoga sessions at a yoga studio compared to participating in online-yoga at home for patients with cancer undergoing oncological treatment. Additionally, the aim is to study health-related outcomes of yoga. Patients diagnosed with cancer undergoing oncological treatment at two hospitals in Sweden will be included in the study. A preference-based allocation will be used, participants chose self if they want to participate in in-person yoga at a studio or in yoga online. Regardless of allocation, the yoga sessions will take place in a group setting once a week for a duration of 12 weeks. All participants will also have access to a yoga application on their tablets or cell phones, with a recommendation to engage in self-guided yoga for at least 10 minutes per day.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cancer and scheduled for or initiated oncological treatment at an oncology clinic.
* Received written information about the study.
* Willing to participate in the study and able to follow the protocol.
* Understanding and expressing themselves in Swedish.
* Age ≥ 18 years.
* Provided informed consent.

Exclusion Criteria:

* Patients with severe cognitive impairments such as dementia and serious psychiatric illness.
* Patients with significant physical disabilities that may hinder yoga.
* Patients with difficulties completing questionnaires.
* Expected survival of less than 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Patients preferences to yoga during oncological treatment | Baseline, 3 months and 6 months
  Interviews on choice of yoga setting: physical or digital

SECONDARY OUTCOMES:
Health-related quality of life | Baseline, 3 months and 6 months
  Health-related quality of life will be assessed by The European Organisation for Research and Treatment of Cancer, Quality of life Questionnaire C30 (EORTC QLQ-C30) which consists of a 30-item questionnaire, covering a global health status/quality of life (QoL) scale, five functioning scales, three symptom scales and six items concerning symptoms. All scales and single-item measures were transformed to scores in the range 0-100. A higher score on the global status scale and the functional scales denotes a high level of health and functioning, while a higher score on the symptomatic scale denotes a high level of symptom burden
Health | Baseline, 3 months and 6 months
  Health will be assessed with EuroQoL which consist of two parts: EuroQoL 5 dimensions 5 levels (EQ 5D 5L) and EuroQoL Visual Analogue Scale (EQ-VAS). EQ-5D 5L comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ-VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'The best health you can image' =100 and 'The worst health you can image' =0.
Anxiety and depression | Baseline, 3 months and 6 months
  The Hospital Anxiety and Depression Scale (HADS) will be used to measure anxiety and depression. The scale consists of 14 items, with seven items related to anxiety and seven related to depression. Each item is scored on a likert scale ranging from 0 to 3, with responses indicating the severity of the symptom from 0=no symptoms to 3= severe symptoms.
Fatigue | Baseline, 3 months and 6 months
  Fatigue will be assessed with the Multidimensional Fatigue Inventory (MFI). The questionnaire consists of 20 items, measuring five subscales of MFI: General, Physical and Mental Fatigue, Reduced Motivation and Reduced Activity. Each item is scored on a likert scale ranging from 1 to 5. Higher scores indicate higher levels of fatigue.
Sleep | Baseline, 3 months and 6 months
  Sleep will be measured with Minimal Insomnia Symptom Scale (MISS). The questionnaire consists of 3 items. Each item is scored on a likert scale ranging from 0 to 4, with responses indicating the severity of the symptom from 0=no symptoms to 5= severe symptoms.
Stress | Baseline, 3 months and 6 months
  Stress will be measured by the questionnaire The Perceived Stress Scale (PSS) which measures general stress and coping capabilities. The instrument has 14 items with 4 alternatives to each item. A higher score indicates higher stress. Each item minimum 0 and maximum 4.
Physical Activity | Baseline, 3 months and 6 months
  Accelerometer
Adherence to the yoga sessions and the application | At 3 months (After completion of the intervention)
  Attendance at yoga-class and time spent (minutes) using the application

CONTACTS AND LOCATIONS:
Overall Officials: Anna Strömberg, PHD, Principal Investigator — Department of Medical and Health sciences, Linköping university, Sweden
Locations (1):
- Department of oncology, university hospital, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No